CLINICAL TRIAL: NCT04266158
Title: Functional Assistance Provided by Myoelectric Elbow-wrist- Hand Orthosis
Brief Title: FAME: Functional Assessment of a Myoelectric Orthosis Hand Orthoses
Acronym: FAME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor stoppage of recruitment
Sponsor: Ohio State University (Other)
Collaborators: Medical University of South Carolina (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016H0339
Record Dates: First submitted 2018-01-10; First posted 2020-02-12 (Actual); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Paresis; Stroke
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- MyoPro 2 Motion-G-orthosis-None (Active Comparator): Following screening, all subjects receive 2 education sessions, during which they are trained on the donning and use of the MyoPro 2 Motion-G, Comfy Splint orthosis, and no device, all on the affected UE. The presentation and training on these interventions is non-randomized and administered to all subjects. After these training sessions, all subjects complete a battery of three tests while wearing one of the two devices, or no device. The order in which the tests are administered is randomized.
  Interventions: Device: Myoelectric UE Device-UE Orthosis-No Device
- Comfy Splint (Active Comparator): Following screening, all subjects receive 2 education sessions, during which they are trained on the donning and use of the MyoPro 2 Motion-G, Comfy Splint orthosis, and no device, all on the affected UE. The presentation and training on these interventions is non-randomized and administered to all subjects. After these training sessions, all subjects complete a battery of three tests while wearing one of the two devices, or no device. The order in which the tests are administered is randomized.
  Interventions: Device: Myoelectric UE Device-UE Orthosis-No Device
- No Splint (Active Comparator): Following screening, all subjects receive 2 education sessions, during which they are trained on the donning and use of the MyoPro 2 Motion-G, Comfy Splint orthosis, and no device, all on the affected UE. The presentation and training on these interventions is non-randomized and administered to all subjects. After these training sessions, all subjects complete a battery of three tests while wearing one of the two devices, or no device. The order in which the tests are administered is randomized.
  Interventions: Device: Myoelectric UE Device-UE Orthosis-No Device

INTERVENTIONS:
Device: Myoelectric UE Device-UE Orthosis-No Device — all subjects receive 2 education sessions, during which they are trained on the donning and use of the MyoPro 2 Motion-G, orthosis, and no device, all on the affected UE. The presentation and training on these interventions is non-randomized and administered to all subjects.

SUMMARY:
The primary study objective is to compare post-stroke upper extremity (UE) movement while wearing a brace called the MyoPro 2 Motion G versus UE movement while wearing a resting splint and no device in stroke survivors with moderate UE dysfunction. During the study, subjects will undergo general training in the operation of the EMG-controlled orthosis and the comparison orthosis, and then guided through a series of standard clinical outcome measures. These outcome measures will allow the researchers to directly compare the relative benefit of the MyoPro 2 Motion G with a resting hand splint and no device in reducing UE impairment and increasing UE dexterity and functional task performance.

ELIGIBILITY:
Inclusion Criteria:

* Manual Muscle Test >1/5 in the paretic biceps, triceps, finger extensors and finger flexors;
* score > 10 < 30 on the Upper extremity Fugl Meyer AND active shoulder flexion of at least 30 degrees with device weight on affected arm;
* Ability to generate consistent, detectable EMG signal from the bicep/tricep upper arm and distal forearm flexor and extensor sensor sites with wrist in neutral, and fingers in neutral. At rest, achieve an EMG of 5 or below on myConfig (wrist and fingers in neutral and elbow extended); with gain at < 10 and boost <12, able to reach a threshold of 10 at both bicep and wrist flexors/extensors;
* a single stroke that is the cause of arm impairment, experienced >12 months ago; if there are additional asymptomatic lesions (as diagnosed by MRI), these subjects may also be included. Those with another symptomatic stroke in addition to the stroke causing arm impairment are excluded;
* score >70 on the Modified Mini Mental Status Examination;
* age >18< 85;
* > 6 months since previous functional or therapeutic use of an upper extremity myoelectric orthosis;
* Height >5'0";
* Weight >110< 250 lbs.;
* Forearm circumference (at widest part) <13 in.;
* Bicep circumference >9 <15 in.;
* Upper arm length >5.5 in.;
* Wrist thickness (anterior- posterior) <1.75 in.;
* ability to stand with minimal assistance

Exclusion Criteria:

* > 5 on a 0-10 Numeric Pain Rating Scale for pain in the paretic hand, arm or shoulder;
* > 3 on the Modified Ashworth Spasticity Scale in the paretic elbow, >2 at wrist or fingers;
* < 2.5 on the Alexander Apraxia scale; '
* history of neurological disorder other than stroke;
* change in anti-spasticity medications in the last 6 months, and/or receipt of botulinum toxin in the paretic UE in the previous 4 months;
* elbow contracture greater than 10 degrees;
* inability to passively extend fingers while wrist is in neutral;
* other conditions or physical/mental attributes that may undermine safety and/or full participation in the study;
* bilateral hemiparesis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Groups:
- 0 - See Description: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Period: Overall Study
Arm/Group | 0 - See Description
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Groups:
- 0 - See Description Below: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.non-randomized and administered to all subjects.
Arm/Group | 0 - See Description Below
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB) — The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: 0 - See Description
Description: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Time Frame: see description above
Population: 0
Groups:
- 0 - See Description Below: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Arm/Group | 0 - See Description Below
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Description: The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.
Arm/Group | 0 - See Description Below
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI is no longer at The Ohio State University and is not actively working at another institution for record transfer. We contacted remaining study team members and department chair to obtain updates for these records. We were told the PI was dismissed and there was alleged noncompliance and misconduct. The study team and department chair are unable to confirm if available documents for these records are accurate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04266158/Prot_000.pdf